CLINICAL TRIAL: NCT03565913
Title: Potential Therapeutic Role of Effervescent Calcium-Magnesium Citrate in Chronic Kidney Disease Stage V
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Henry Quinones, Professor, Internal Medicine - Nephrology, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU 122016-001
Record Dates: First submitted 2018-05-18; First posted 2018-06-21 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: CKD Stage 5
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — effervescent calcium magnesium citrate; Solutions

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized into two groups in a parallel design. One group will take EffCaMgCit 15 meq (300 mg) Ca, 10 meq Mg (122 mg) and 45 meq total citrate thrice daily, while the other group will take calcium acetate suspension/solution (CaAcS) 15 meq Ca thrice daily for two years.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: To provide adequate blinding, each medication sachet will be labelled with the study name, IRB number, principal investigator's name, expiration date and identification number of the study subject. Labels will be applied to the appropriate medication sachets once the subject has been randomized and assigned to a treatment group. Labelling of the sachets will be done by non-patient care personnel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- EffCaMgCit (Experimental): Patients in the EffCaMgCit group will receive 45 meq (900 mg) Ca, 30 meq (365 mg) Mg, and 135 meq total citrate per day from 3 months to 2 years.
  Interventions: Drug: EffCaMgCit
- CaAcS (Active Comparator): Patients in the CaAcS group will take 45 meq (900 mg) Ca and 45 meq acetate (without Mg or citrate) per day.
  Interventions: Other: CaAcS

INTERVENTIONS:
Drug: EffCaMgCit — Patients in the EffCaMgCit group will receive 45 meq (900 mg) Ca, 30 meq (365 mg) Mg, and 135 meq total citrate per day from 3 months to 2 years.
  Other Names: Effervescent calcium magnesium citrate
  Arms: EffCaMgCit
Other: CaAcS — CaAcS group will take 45 meq (900 mg) Ca and 45 meq acetate (without Mg or citrate), three times daily for 2 years
  Other Names: Calcium acetate suspension/solution
  Arms: CaAcS

SUMMARY:
The Investigators plan to conduct a long-term trial to explore therapeutic implications of effervescent calcium magnesium citrate (EffCaMgCit) in CKD Stage V (end stage renal disease on hemodialysis). The Investigators will test the hypothesis that EffCaMgCit would retard the formation of calciprotein particles (CPP) in CKD Stage V, thereby reducing the degree of coronary artery and peripheral artery calcification and cardiac hypertrophy-fibrosis.

Aim 1. To compare cardiovascular risk of EffCaMgCit versus CaAcS in CKD Stage V Aim 2. To show that EffCaMgCit reduces putative serum FGF23, and increases beneficial alkali load Aim 3. To compare parameters of bone turnover and bone mineral density (BMD) between EffCaMgCit and CaAcS groups

DETAILED DESCRIPTION:
150 adult subjects (> 21 years of age, any cause of CKD) of either gender of any ethnicity with CKD Stage V on hemodialysis will be recruited from Davita-UTSW dialysis centers and randomized into two equal groups in a parallel design, stratified according to gender and age (> or ≤ 50 years). After baseline evaluation, one group (EffCaMgCit Group) will take EffCaMgCit, and the other group (CaAcS Group) will take calcium acetate suspension/solution for two years. Both drugs will be taken 1 sachet each just before or along with breakfast and dinner for the first three months. If tolerated, the dose will be increased to 1 sachet tid just before or along with breakfast, lunch and dinner.

After screening and a baseline evaluation, research personnel will visit patients at the dialysis center every three months for two years. Patients will be evaluated with a medical history, side effect questionnaires, blood pressure measurements, blood tests, echocardiograms, coronary artery calcification analyses, muscle magnesium analyses, and bone mineral density analyses.

It is expected that markers of cardiovascular risk would be improved in patients taking CaMgCit, and would remain stable in those taking CaAcS.

Endpoint Expectations:

* During treatment with EffCaMgCit, T50 would increase (indicative of reduced propensity for CPP formation)
* Serum Mg (inhibitor of CPP formation) would be increased by EffCaMgCit
* An increase in intracellular muscle Mg would show that EffCaMgCit provides a Mg load, and also indicates repletion of Mg stores that might be cardioprotective independently of effects on CPP formation
* The Investigators anticipate that serum FGF23 would be lower and serum Klotho would be higher on EffCaMgCit

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (> 21 years of age, any cause of CKD) of either gender of any ethnicity with CKD Stage V on hemodialysis will be recruited. Patients with Type II diabetes and hypertension will be allowed. Treatment with drugs for management of osteoporosis (bisphosphonate, teriparatide, or denosumab) or for chronic kidney disease, customary drugs for hypertension or diabetes, and exogenous estrogen or selective estrogen receptor modulators will be allowed.

Exclusion Criteria:

* Patients with serum Mg > 3.65 mg/dL (3 meq/L) will be excluded (de Francisco, 2010). Also excluded from the study will be those with bowel disease, hypercalcemia, hypophosphatemia (serum P < 2.5 mg/dL) and treatment with adrenocorticosteroids or aluminum-containing antacids or drugs.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2017-01-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum T50 for CPP | 24 months
  The maturation time (T50) of calciprotein particles in serum will be measured. T50 CPP (measured by Calcisco using Pasch's method) assays the kinetics of transformation from primary to secondary CPP in vitro. Fresh serum samples will be kept at -80 degrees until shipment to Calcisco AG (Berne, Switzerland) for T50 analysis, which will determine T50 of CPP through research collaboration with CMMCR.

SECONDARY OUTCOMES:
Intracellular muscle magnesium | 24 months
  Intracellular Mg will be measured in calf muscle, by using 31P magnetic resonance spectroscopy, based on the formula: [Mg] - kd(10.796-D)/(D-8.251), in which kd is the dissociation constant for MgATP complex (=50 µM) and D is the chemical shift difference between alpha- and beta-ATP 31P signals observed in 31P MR spectrum.
Control of hyperphosphatemia and serum FGF23 | 24 months
  The control of hyperphosphatemia will be evaluated from changes in serum P concentration, serum FGF23 and Klotho.
Parathyroid function and bone turnover | 24 months
  Parathyroid function will be evaluated from serum PTH, vitamin D status from serum calcitriol, bone resorption from serum CTX, and bone formation from serum BSAP. Change in bone mass will be evaluated by BMD (proximal femur, L2-L4 spine and distal third of radius).

CONTACTS AND LOCATIONS:
Overall Officials: Henry Quinones, MD, Principal Investigator — UTSW
Locations (1):
- DaVita Dialysis Centers, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided